CLINICAL TRIAL: NCT04253899
Title: The Management of Perforated Acute Appendicitis: A Randomized Control Trial in the Adult and Pediatric Populations
Brief Title: The Management of Perforated Acute Appendicitis in Adult and Pediatric Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Juan Sanabria, Professor of Surgery, Marshall University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504002-3
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Perforated Appendicitis
Keywords: Perforated appendicitis; Pediatric appendicitis; Appendectomy; Appendiceal abscess; Antibiotic Therapy
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard pediatric group: (Active Comparator): patients ≤17 yo with acute perforated appendicitis and interval appendectomy (n=25)
  Interventions: Procedure: Appendectomy
- Experimental pediatric group: (Experimental): patients ≤17 yo with acute perforated appendicitis abscess and observation (n=25)
  Interventions: Other: Observation
- Standard adult group: (Active Comparator): patients ≥18 yo with acute perforated appendicitis and interval appendectomy (n=25)
  Interventions: Procedure: Appendectomy
- Experimental adult group: (Experimental): Patients ≥18 yo with acute perforated appendicitis and observation (n=25)
  Interventions: Other: Observation

INTERVENTIONS:
Procedure: Appendectomy — Interval Appendectomy
  Arms: Standard adult group:; Standard pediatric group:
Other: Observation — observation and follow up
  Arms: Experimental adult group:; Experimental pediatric group:

SUMMARY:
Patients admitted at Marshall Health - Cabell Huntington Hospital with the diagnosis of acute perforated appendicitis or appendicular abscess larger than 3cm will be admitted and treated with percutaneous drainage and the IV antibiotics for 3 days. If the patient becomes afebrile and has a normal WBC, the patient will stay in the hospital for a single day with oral antibiotics and then will be discharged to continue oral antibiotics for seven more days. If the patient is febrile or has elevated WBC either after the 3 days of IV antibiotics or the single day of oral antibiotics, the patient will complete a course of IV antibiotics for a total of seven days. If still febrile, the patient will undergo further assessment.

A follow up will be conducted ~10 days after discharge from the hospital to determine if the patient is still symptomatic or asymptomatic. Asymptomatic patients will be followed up every month for 3 months, while symptomatic patients will be treated as needed. After 12 weeks, subjects will be randomized to interval appendectomy vs observation. Follow-ups will occur every 3 months for 12 months, when the study will be concluded.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all ages.
* Clinical and radiological diagnosis by contrast CT scan of acute perforated appendicitis.
* Formal consent for the present study must be signed by the patient or his/her parents
* Patients with initial presentation of a phlegmon (abscess in evolution)

Exclusion Criteria:

* Patients with non-perforated appendicitis
* Presentation with initially non-perforated appendicitis but found perforation at surgery
* Patient with septic shock
* Patients who had previous appendectomy
* Current treatment of malignancy
* Immunocompromised patients
* Positive pregnancy test
* No consent for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Determine rate and severity of complications after interval appendectomy | 12 months
Determine the incidence and rate of appendectomies (in the observation arm) during the first year of diagnosis | 12 months

SECONDARY OUTCOMES:
Determine the rate of complete response after percutaneous drainage and antibiotic therapy | 12 months
Determine the mean surgical value (quality/cost) for each group | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanabria, MD MSc FACS, Principal Investigator — Marshall University School of Medicine
Locations (1):
- Marshall University School of Medicine, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No